CLINICAL TRIAL: NCT04684758
Title: HIV Acquisition and Life Course of Born-abroad Men Who Have Sex With Men Living in Ile-de-France: the GANYMEDE Study
Acronym: GANYMEDE
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 14058
Record Dates: First submitted 2020-12-03; First posted 2020-12-28 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Men Who Have Sex With Men; People Living With HIV
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-completion of a questionnaire — The questionnaire will be translated into 5 languages (English, Spanish, Portuguese, Arabic, and Russian) in order to allow almost all of the participants to answer the survey themselves, without assistance. In order to not exclude those who cannot read, or those who do not master any of the 6 languages offered, the questionnaire may be administered with the assistance of a member of the research team of the associated center, including through a telephone interpretation service, if necessary.

SUMMARY:
In France, men who have sex with men (MSM) born abroad are the most affected population by HIV, in terms of HIV incidence and prevalence of undiagnosed infections. Close to 50% of born-abroad HIV-infected MSM are living in the region of Ile-de-France, which is the metropolitan area of Paris. Recent European data, not including France, suggest that born-abroad MSM have the highest rate of post-migration HIV acquisition. Many vulnerability factors could explain le burden of HIV in this group of the population.

A better understanding of vulnerability factors related to post-migration HIV acquisition should allow to improve HIV prevention and screening strategies among born-abroad MSM living in France. This, in turn, should reduce the burden of HIV in this population in France.

DETAILED DESCRIPTION:
A better understanding of vulnerability factors related to post-migration HIV acquisition should allow to improve HIV prevention and screening strategies among born-abroad MSM living in France. This, in turn, should reduce the burden of HIV in this population in France.

Multicenter, cross-sectional, two-year study in the region Ile-de-France. The study is based on the self-completion of a questionnaire, built after an exploratory qualitative study.

Constitution of a representative sample of born-abroad HIV-infected MSM from patients followed up for HIV in Paris area. Questionnaires will collect data needed to estimate the post-migration HIV acquisition rates, and will explore contextual and individual factors leading to high exposure to HIV.

The participants will complete a questionnaire translated into 5 languages (English, Spanish, Portuguese, Arabic, and Russian) in order to allow almost all of the participants to answer the survey themselves, without assistance. In order to not exclude those who cannot read, or those who do not master any of the 6 languages offered, the questionnaire may be administered with the assistance of a member of the research team of the associated center, including through a telephone interpretation service. A brief eCRF will collect clinical and biological data, and historical viral sequences in associated virology departments, when available.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gender men who report having sex with men;
* Over 18 years of age;
* Type 1 HIV infected;
* Born in a country other than France and arrived in France at the age of 15 at the earliest;
* Followed in Ile-de-France for their HIV infection and having consulted at least once in the participating center during the last 12 months;
* Non-opposition to the collection of their health data, after being well informed of the study and the patient rights in accordance with RGPD and LIL (French regulation)

Exclusion Criteria:

* Somatic or psychiatric pathology making it impossible to participate in an investigation;
* Communication disorder making it impossible to read (or oral responses in the event of assisted questionnaire completion).

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Cis-gender men who report having sex with men;
  * Over 18 years of age;
  * Type 1 HIV infected;
  * Born in a country other than France and arrived in France at the age of 15 at the earliest;
Sampling Method: Non-Probability Sample
Enrollment: 1048 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Post-migration proportion of HIV acquisition in born-abroad HIV-positive MSM living in Ile-de-France | Through study completion, an average of 12 months
  Estimation of the post-migration proportion of HIV acquisition in born-abroad HIV-positive MSM living in Ile-de-France (proportion of participants, n (%))

SECONDARY OUTCOMES:
Timing of HIV infection for people infected in France | Through study completion, an average of 12 months
  Estimation of the timing of HIV infection for people infected in France (years, median, IQR)

OTHER OUTCOMES:
Phylogenetic analysis in participants having acquired HIV before and after the migration, between them and with other populations | Through study completion, an average of 12 months
  Comparing the viral sequence from participant samples, will allow to estimate the proportion of viral sequences included in viral clusters comprising viral sequences from patients born in France and born outside France (proportion of participants, n (%))
Motivations and migratory processes | Through study completion, an average of 12 months
  Analyses of participant questionnaires, will identify the motivations and the migratory processes in the global context of the country of origin (proportion of participants per item, based on responses to questionnaire, n (%))
Vulnerability factors | Through study completion, an average of 12 months
  To determine the vulnerability factors for HIV infection, including social inequalities in health, in the country of origin, during the migration, and in France (proportion of participants per item, based on responses to questionnaire, n (%))
Health contacts | Through study completion, an average of 12 months
  Description of health contacts, if any, with health system before HIV diagnosis (proportion of participants per item, based on responses to questionnaire (%))
Missed opportunities of pre-exposure prophylaxis | Through study completion, an average of 12 months
  Description of missed opportunities of pre-exposure prophylaxis access (proportion of participants per item, based on responses to questionnaire, n (%))
HIV healthcare | Through study completion, an average of 12 months
  Description of HIV care, including antiretroviral treatment and viral suppression coverage (proportion of participants, n (%))

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié-Salpêtrière, AP-HP, Institut Pierre Louis d'Épidémiologie et de Santé Publique (iPLESP), INSERM 1136, Paris, France

IPD SHARING:
Plan to Share IPD: No